CLINICAL TRIAL: NCT04667611
Title: Patient-reported Outcome Measures (PROMs) as Characteristics and Prognostic Factors in Patients With Bodily Stress Syndrome: Protocol for a Prospective Cohort Study
Brief Title: Patient-reported Outcome Measures (PROMs) in Patients With Bodily Stress Syndrome: Protocol for a Prospective Cohort Study
Acronym: SYMPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Helena Liira, Chief Physician, Helsinki University Central Hospital
Other Study IDs: 1159007
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Somatic Symptom; Chronic Fatigue Syndrome; Fatigue; Dysphagia; Exhaustion; Syndrome
Keywords: bodily stress syndrome; functional somatic symptoms; functional somatic syndrome
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Medically Unexplained Symptoms; Fatigue Syndrome, Chronic; Fatigue; Deglutition Disorders; Syndrome | interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild
  Interventions: Behavioral: Psychosocial interventions
- Moderate
  Interventions: Behavioral: Psychosocial interventions
- Severe
  Interventions: Behavioral: Psychosocial interventions

INTERVENTIONS:
Behavioral: Psychosocial interventions — Cognitive behavioural therapy (CBT) based individual and group intervention

SUMMARY:
This cohort study implements patient reported outcome measures (PROMs) for patients with bodily stress syndrome in a clinic for functional disorders.

DETAILED DESCRIPTION:
The Sympa Cohort study is a prospective, single site cohort study that consists of administration of PROMs questionnaires to patients that attend the Clinic for Functional Disorders at Helsinki University hospital (HUS). The questionnaires are handed out to the study population within seven days before their first visit at the clinic, and then at the following 3, 6 and 12 months. The study population consists of consecutive adult patients that are referred to the clinic either from other hospital units or primary care. The collected data will later be linked with national registries on diagnoses, medication use and work ability. The Sympa Cohort study may have implications in targeting the factors influencing functional outcomes and quality of life reported by patients with bodily stress syndrome. It will also form a quality register for the Clinic and characterize the first systematic collection of PROMs related to these disorders in Finland.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* Age 18-80 years
* Referred to Clinic for Functional Disorders either from other hospital units or from primary care
* Willingness to be enrolled in the study, by signing the informed consent

Exclusion Criteria:

* Patients not able to fill in the forms in Finnish or due to physical constraints (e.g. dystonia)
* Symptoms are likely due to a somatic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive patients referred to the Clinic for Functional Disorders and who give their consent to be followed up during one year after their visit to the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Self-rated global health improvement | 12 months
  Measured by clinical improvement scale (clinical global improvement, CGI), a five-point Likert scale
Functional ability | 12 months
  Measured by WHODAS 2.0

SECONDARY OUTCOMES:
PHQ-9 | 3, 6 and 12 months
  Depression
GAD-7 | 3, 6 and 12 months
  Anxiety
EUROHIS-QOL-8 | 3, 6 and 12 months
  Health related quality of life
15D | 3, 6 and 12 months
  Health related quality of life
SSD-12 | 3, 6 and 12 months
  Symptom severity
RS-14 | 3, 6 and 12 months
  Resilience

CONTACTS AND LOCATIONS:
Overall Officials: Helena Liira, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Clinic for Functional Disorders, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No